CLINICAL TRIAL: NCT01214486
Title: Measurement of Plasma and Intracellular Concentrations of Raltegravir in Patients Infected With Human Immunodeficiency Virus
Brief Title: Measurement of Plasma and Intracellular Concentrations of Raltegravir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Principal Investigator, Uriel Sandkovsky, MD, Principal Investigator, University of Nebraska
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 506-10-FB
Record Dates: First submitted 2010-09-28; First posted 2010-10-05 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: HIV
Keywords: HIV; RAL; Raltegravir; Isentress; Pharmacokinetics
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Subjects should be on RAL 400mg twice daily at least 1 week. Subjects will be asked to come to the Specialty Clinic at two different points on the same day: at either 2, 4 or 6 hours after taking the drug, and at 10 or 12 hours after taking the drug. After completion of the first part of the study, subjects whose viral load is below the limit of detection (HIV RNA < 50 copies/mL) will be asked to switch to once a day RAL dosing (i.e. 800 mg once a day). Once the a subject has taken RAL once a day for at least three consecutive days, s/he will be asked to come to the Specialty Clinic at two different points in the same day to obtain blood by venous puncture. Blood will be obtained 2 or 4 hours after the dose and at 20-24 hours after the dose.
  Other Names: RAL; Isentress

SUMMARY:
The primary purpose of this study is to analyze and compare plasma and intracellular concentrations of Raltegravir (RAL) in blood plasma and in peripheral blood mononuclear cells, using high performance liquid chromatography (HPLC).

DETAILED DESCRIPTION:
Integrase strand transfer inhibitors are one of the newest class of antiretroviral drugs. This class of drugs inhibit the catalytic activity of HIV-1 integrase, an HIV-1-encoded enzyme required for viral replication [1]. Inhibition of integrase prevents covalent insertion of unintegrated, linear HIV-1 DNA into the host cell genome, therefore preventing the formation of HIV-1 provirus. RAL, the first agent in its class, was initially approved in 2007 for use in patients harboring drug-resistant HIV [2]. More recently, the FDA has expanded the indication for RAL use in HIV-infected patients who are antiretroviral naïve [3]. The currently approved dose is 400 mg twice daily. The RAL area-under-the-curve (AUC) and Cmax increase in a dose-dependent fashion over the range of 100 mg to 1,600 mg. With twice-daily dosing, PK steady state is achieved within approximately the first 2 days. Considerable variability was observed in the PK of raltegravir in clinical trials. In clinical trial participants receiving twice-daily RAL 400 mg, drug exposures were characterized by a geometric mean AUC within the first 12 hours of 14.3 mcM(hr) and a plasma concentration at 12 hours of 142 nM [3]. RAL at concentrations of 6 to 50 nM resulted in 95% inhibition (EC95) of viral spread in mitogen-activated human peripheral blood mononuclear cells (PBMCs) infected with diverse, primary clinical isolates of HIV-1, including isolates resistant to reverse transcriptase inhibitors and protease inhibitors (PIs).

The absolute bioavailability of RAL has not been established. RAL is approximately 83% bound to human plasma protein over the concentration range of 2 to 10 mcM. The apparent terminal half-life of RAL is approximately 9 hours, with a shorter alpha-phase half-life (about 1 hour), accounting for much of the AUC. Determination of drug levels to guide treatment of HIV infection is available for protease inhibitors (PI) and non-nucleoside reverse transcriptase inhibitors (NNRTI) but is not yet considered standard of care [4,5]. RAL is associated with potent performance against HIV in treatment-naïve patients and those with limited treatment options, potentially because of its binding interaction with the HIV preintegration complex. When RAL binds to the complex, the drug dissociates at a rate slower than the half-life of the complex itself, which makes binding essentially irreversible. Thus, the efficacy of RAL may be dependent on intracellular binding levels of the drug to the preintegration complex, rather than on the plasma concentrations of RAL. Because of this, we postulate that intracellular concentrations of RAL are more likely to correlate with biological activity against HIV. Moreover, if pharmacokinetic behavior can be predicted, and depending on the trough concentrations observed, the drug might be suitable for different dosing approaches including once a day administration. This would create more flexibility for patients, and the chance to improve adherence.

ELIGIBILITY:
Inclusion Criteria:

* Be of age greater than or equal to 19 years
* Have documented HIV
* Be taking RAL for at least 7 days

Exclusion Criteria:

* Any acute intercurrent illness that might interfere with the interpretation of the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2011-04-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Concentrations of RAL in blood cells. | one month
  Analyze and compare plasma and intracellular concentrations of RAL in blood plasma and in peripheral blood mononuclear cells, using high performance liquid chromatography (HPLC).
Concentrations of RAL in blood plasma. | one month
  Analyze and compare plasma and intracellular concentrations of RAL in blood plasma and in peripheral blood mononuclear cells, using high performance liquid chromatography (HPLC).

SECONDARY OUTCOMES:
Pharmacokinetic variability of plasma concentrations of the drug. | one month
  To determine the pharmacokinetic variability of plasma and intracellular concentrations of the drug.
Pharmacokinetic variability of intracellular concentrations of the drug. | one month
  To determine the pharmacokinetic variability of plasma and intracellular concentrations of the drug.
Trough concentrations of the drug when dosed twice daily versus once daily. | one month
  To compare pharmacokinetics of the drug when dosed twice daily versus once daily.
Pharmacokinetics of the drug when dosed twice daily versus once daily. | One month
  To compare pharmacokinetics of the drug when dosed twice daily versus once daily.

CONTACTS AND LOCATIONS:
Overall Officials: Uriel S Sandkovsky, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Thompson MA, Aberg JA, Cahn P, Montaner JS, Rizzardini G, Telenti A, Gatell JM, Gunthard HF, Hammer SM, Hirsch MS, Jacobsen DM, Reiss P, Richman DD, Volberding PA, Yeni P, Schooley RT; International AIDS Society-USA. Antiretroviral treatment of adult HIV infection: 2010 recommendations of the International AIDS Society-USA panel. JAMA. 2010 Jul 21;304(3):321-33. doi: 10.1001/jama.2010.1004. PMID 20639566
- [Background] Hicks C, Gulick RM. Raltegravir: the first HIV type 1 integrase inhibitor. Clin Infect Dis. 2009 Apr 1;48(7):931-9. doi: 10.1086/597290. PMID 19231980
- [Background] 3. http://www.merck.com/product/usa/pi_circulars/i/isentress/isentress_pi.pdf
- [Background] de Maat MM, Huitema AD, Mulder JW, Meenhorst PL, van Gorp EC, Mairuhu AT, Beijnen JH. Subtherapeutic antiretroviral plasma concentrations in routine clinical outpatient HIV care. Ther Drug Monit. 2003 Jun;25(3):367-73. doi: 10.1097/00007691-200306000-00018. PMID 12766566
- [Background] Powderly WG, Saag MS, Chapman S, Yu G, Quart B, Clendeninn NJ. Predictors of optimal virological response to potent antiretroviral therapy. AIDS. 1999 Oct 1;13(14):1873-80. doi: 10.1097/00002030-199910010-00009. PMID 10513645
- [Background] Shah VP, Midha KK, Findlay JW, Hill HM, Hulse JD, McGilveray IJ, McKay G, Miller KJ, Patnaik RN, Powell ML, Tonelli A, Viswanathan CT, Yacobi A. Bioanalytical method validation--a revisit with a decade of progress. Pharm Res. 2000 Dec;17(12):1551-7. doi: 10.1023/a:1007669411738. No abstract available. PMID 11303967
- [Background] Viswanathan CT, Bansal S, Booth B, DeStefano AJ, Rose MJ, Sailstad J, Shah VP, Skelly JP, Swann PG, Weiner R. Quantitative bioanalytical methods validation and implementation: best practices for chromatographic and ligand binding assays. Pharm Res. 2007 Oct;24(10):1962-73. doi: 10.1007/s11095-007-9291-7. Epub 2007 Apr 26. PMID 17458684
- [Background] King T, Bushman L, Anderson PL, Delahunty T, Ray M, Fletcher CV. Quantitation of zidovudine triphosphate concentrations from human peripheral blood mononuclear cells by anion exchange solid phase extraction and liquid chromatography-tandem mass spectroscopy; an indirect quantitation methodology. J Chromatogr B Analyt Technol Biomed Life Sci. 2006 Feb 2;831(1-2):248-57. doi: 10.1016/j.jchromb.2005.12.033. Epub 2006 Jan 10. PMID 16412710
- [Background] Remmel RP, Kawle SP, Weller D, Fletcher CV. Simultaneous HPLC assay for quantification of indinavir, nelfinavir, ritonavir, and saquinavir in human plasma. Clin Chem. 2000 Jan;46(1):73-81. PMID 10620574
- See also: University of Nebraska Medical Center HIV Clinic — http://www.unmc.edu/hiv